CLINICAL TRIAL: NCT01315964
Title: Effects of Dietary Plant Stanol Esters of Blood Flow Among Healthy Adult Human Subject. The BLOOD FLOW -Study
Brief Title: Effects of Plant Stanol Esters on Blood Flow
Acronym: BLOOD FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Institute of Occupational Health (Other)
Responsible Party: Principal Investigator, Markku Nissinen, MD PhD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3352
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Atherosclerosis
Keywords: cholesterol; plant sterols; atherosclerosis; arterial stiffness
MeSH Terms: conditions — Atherosclerosis | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- plant stanol ester (Active Comparator): 3 grams of plant stanol esters per day in a margarine product as part of daily diet for 6 months
  Interventions: Dietary Supplement: plant stanol ester
- Placebo (Placebo Comparator): a margarine product as part of daily diet, which is not containing plant stanol esters
  Interventions: Dietary Supplement: plant stanol ester

INTERVENTIONS:
Dietary Supplement: plant stanol ester — 3 gr of plant stanol esters per day in a margarine product as part of daily diet for a period of 6 months
  Other Names: Benecol

SUMMARY:
Plant stanol esters as part of daily diet can decrease serum level of LDL-cholesterol up to 10%. This decrease diminishes the risk of development of premature atherosclerosis and it´s complications (e.g., acute myocardial infarction) in adult human subjects.

The purpose of the present study is to evaluate among healthy human subjects (N=100) effects of plant stanol esters (3 grams/day for 6 months) as part of daily diet in margarine on arterial endothelial cells, arterial stiffness, autonomic innervation of the arteries, arterial blood flow and serum fats. The non-invasive arterial measurements (VaSera®, EndoPat® and WinCRPS®) are performed and blood samples are taken at the beginning and at the end of the 6-month-long study period. Also questionnaires concerning healthy, and life and dietary habits are fulfilled. Dietary records (twice for a 3-day-period) are done.

Hypothesis of the study is that a dietary serum cholesterol lowering intervention has beneficial influence on the early prognostic markers of premature atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* healthy human subjects

Exclusion Criteria:

* abnormal liver, kidney and thyroid function
* unstable myocardial disease
* inflammatory bowel disease
* alcohol abuse
* pregnancy
* any lipid-lowering medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Structure and function of the arterial wall | 6 months

SECONDARY OUTCOMES:
serum composition of fats | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Markku J Nissinen, MD Docent, Study Director — Dept. of Medicine, Div. of Gastroenterology, Helsinki Univ. Central Hospital
Locations (1):
- Biomedicum Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Ruuth M, Aikas L, Tigistu-Sahle F, Kakela R, Lindholm H, Simonen P, Kovanen PT, Gylling H, Oorni K. Plant Stanol Esters Reduce LDL (Low-Density Lipoprotein) Aggregation by Altering LDL Surface Lipids: The BLOOD FLOW Randomized Intervention Study. Arterioscler Thromb Vasc Biol. 2020 Sep;40(9):2310-2321. doi: 10.1161/ATVBAHA.120.314329. Epub 2020 Jul 2. PMID 32611242
- [Derived] Hallikainen M, Halonen J, Konttinen J, Lindholm H, Simonen P, Nissinen MJ, Gylling H. Diet and cardiovascular health in asymptomatic normo- and mildly-to-moderately hypercholesterolemic participants - baseline data from the BLOOD FLOW intervention study. Nutr Metab (Lond). 2013 Oct 7;10(1):62. doi: 10.1186/1743-7075-10-62. PMID 24499098
- [Derived] Gylling H, Halonen J, Lindholm H, Konttinen J, Simonen P, Nissinen MJ, Savolainen A, Talvi A, Hallikainen M. The effects of plant stanol ester consumption on arterial stiffness and endothelial function in adults: a randomised controlled clinical trial. BMC Cardiovasc Disord. 2013 Jul 10;13:50. doi: 10.1186/1471-2261-13-50. PMID 23841572